CLINICAL TRIAL: NCT01564602
Title: Prospective Cohort Study to Compare to 2-channel and Multiple Channel Single Port Laparoscopic-assisted Vaginal Hysterectomy
Brief Title: To Compare to 2-channel and Multiple-channel Single Port Laparoscopic-assisted Vaginal Hysterectomy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Taipei Veterans General Hospital, Taiwan (Other Government)
Responsible Party: Principal Investigator, vghtpe user, Director, Taipei Veterans General Hospital, Taiwan
Allocation: Not Applicable | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: VGH2011-03-011IA
Record Dates: First submitted 2012-02-20; First posted 2012-03-28 (Estimated); Last update posted 2012-04-02 (Estimated); Status verified 2012-03

CONDITIONS: Myoma; Adenomyosis
Keywords: 2-channel single port laparoscopy; multiple-channel port laparoscopy
MeSH Terms: conditions — Myoma; Adenomyosis

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (1):
- single port laparoscopic surgery (Experimental): 2-channel or multiple channel single port laparoscopic surgery in gynecologic disorders
  Interventions: Device: comparison multiple channel port laparoscopic surgery

INTERVENTIONS:
Device: comparison multiple channel port laparoscopic surgery — to compare 2-channel single port and multiple channel port laparoscopic surgery
  Other Names: multiple channel port laparoscopic surgery

SUMMARY:
The main objective of this trial is to assess the efficacy and safety of single port-access laparoscopic-assisted vaginal hysterectomy. The operative time, weight of the uterus, blood loss and hospital stay will be record, respectively. The pain score is based on the visual analogue scale in which patients record the intensity of their pain 12, 24, and 48 hours after surgery.

DETAILED DESCRIPTION:
Single port laparoscopy is an attempt to further enhance the cosmetic benefits of minimally invasive surgery while minimizing the potential morbidity associated with multiple incisions. Preliminary advances in LESS as applied to urologic and gastrointestinal surgery demonstrate that the techniques are feasible provided that both optimal surgical technical expertise with advanced skills and optimal instrumentation are available. Recently, Lee et al. performed the multiple channel single port-access laparoscopic-assisted vaginal hysterectomy (SPA-LAVH) in 24 patient. All cases but 3 were performed exclusively through a single port. The median operative time, weight of the uterus, and estimated blood loss were 119 minutes (range 90 to 255 minutes), 347 g (range 225 to 732 g), and 400 mL (range 100 to 1000 mL), respectively. The median hospital stay (postoperative day) was 3 days (range 3 to 7). Although there are a limited number of studies demonstrating the feasibility of single-port access laparoscopic-assisted vaginal hysterectomy (LAVH), single-port surgery is "new-old" (i.e., a revisited and unstandardized technique) because the major disadvantage of limited movement caused by collisions of the laparoscopic instruments has been mitigated by the development of multi-channel approaches. Therefore, the investigators used a 2-channel single-port system, which was different from the previously published 3-channel single-port technique11,12 to reduce collisions and aid the assistant in controlling the scope without interfering with the surgeon's instruments. To our knowledge, there are no randomize control trial to evaluate of 2-channel or multiple channel single port laparoscopic surgery in gynecologic disorders. The purpose of this study was to assess the feasibility of 2-channel and multiple-channel single port laparoscopy in the treatment of benign uterine disease.

ELIGIBILITY:
Inclusion Criteria:

* Patients receive laparoscopic-assisted vaginal hysterectomy (LAVH)
* American Society of Anesthesiologists (ASA) physical status of patient: classification I-II

Exclusion Criteria:

* The procedure will be required to conversion to laparotomy.
* Any cardio-vascular diseases.
* Malignant disease

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2011-01; Primary Completion 2014-01 (Estimated); Study Completion 2014-12 (Estimated)

PRIMARY OUTCOMES:
The operative time | We will follow the patients until one month after the surgery.
  We will follow the patients until one month after the surgery. The primary outcome measure of this trial is the effect and safety of single port-access laparoscopic-assisted vaginal hysterectomy.

SECONDARY OUTCOMES:
weight of the uterus | one month
blood loss | one month
hospital length of stay | one month
morbidity | one month

CONTACTS AND LOCATIONS:
Overall Officials: Yi-Jen Chen, PHD, Study Director — Taipei Veterans General Hospital, Taiwan
Locations (1):
- Taipei Veterans General Hospital, Taipei, Taiwan